CLINICAL TRIAL: NCT05490251
Title: Biological Pathways in Stress Reactivity and Nicotine Addiction Among African American and White Smokers
Brief Title: Translational Research Center in Lung Cancer Disparities (TRACER) Project 2
Acronym: TRACER
Status: Completed | Type: Observational
Sponsor: Virginia Commonwealth University (Other)
Collaborators: City of Hope Medical Center (Other); Medical University of South Carolina (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: MCC-21-18891; 00116801 (Other: Medical University of South Carolina); HM20022956 (Other: Virginia Commonwealth University)
Record Dates: First submitted 2022-05-05; First posted 2022-08-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Smoking; Smoking Behaviors; Smoking Cessation; Stress Reaction
MeSH Terms: conditions — Smoking; Smoking Cessation; Fractures, Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Saliva will be conducted for analyzing biomarkers of stress (i.e. cortisol, alpha-amylase), and biomarkers related to smoking (i.e. cotinine)
  Urine will be collected to determine the presence of illicit substances as an indicator of exclusion/inclusion into the study.
  Patients that provide consent will have additional saliva and urine collected and stored in a centralized biorepository for future research
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to examine racial differences in smoking behaviors and stress responses between African American and white male smokers.

DETAILED DESCRIPTION:
Cigarette smoking is a leading cause of morbidity and mortality from lung cancer among adults in the US. Stress relief and smoking cessation is the best preventive strategy for reducing lung cancer risk and addressing racial disparities in outcomes. Despite this, racial differences are found among those that make quit attempts. Stress has been found to be related to smoking initiation, maintenance, and relapse. Yet, differences in stress responses have not been examined between African American and white smokers. Therefore, this study will examine racial differences in stress responses and smoking behaviors between African American and white male smokers

ELIGIBILITY:
Inclusion Criteria:

* African American and white males
* Between the ages of 18-75 years old
* Smoke at least 5 to 10 cigarettes per day

Exclusion Criteria:

* Smokers who have a serious cognitive disorder
* Have a personal history of lung cancer
* Personal history of usage of illicit drug and alcohol abuse
* Enrollment in a smoking cessation treatment program during the past 6 months
* Current use of a nicotine replacement therapy
* Have any positive responses on the Mini International Neuropsychiatric Interview (MINI) screener

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: African American and white male daily smokers who are between the ages of 18-75 and who smoke at least 5 to 10 cigarettes per day.
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2024-01-31 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Examining racial differences in acute stress responses | Within 1 month following baseline
  Examine racial differences in acute stress responses using a validated psychological stress challenge called the Trier Social Stress Test (TSST)
Examining changes in daily cortisol patterns according to race | Baseline, 4- and 8 weeks post Trier Social Stress Test laboratory visit
  Examine racial differences in daily diurnal cortisol slopes to evaluate hypothalamic-pituitary-adrenal-axis dysregulation and acute stress
Examine changes in stress responses and smoking behaviors as it relates to social determinant factors | Baseline, 4- and 8-weeks post Trier Social Stress Test laboratory visit
  Patients will be administered a survey using validated measures to examine socioeconomic, structural, and psychosocial stressors that impact daily stress and smoking behaviors

CONTACTS AND LOCATIONS:
Overall Officials: Robert Winn, MD, Principal Investigator — Virginia Commonwealth University
Locations (2):
- United States (2):
  - University of Southern California, Los Angeles, California
  - Medical University of South Carolina, Charleston, South Carolina

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-11-09): https://cdn.clinicaltrials.gov/large-docs/51/NCT05490251/Prot_SAP_000.pdf
  • Informed Consent Form (2021-11-29): https://cdn.clinicaltrials.gov/large-docs/51/NCT05490251/ICF_001.pdf